CLINICAL TRIAL: NCT02274467
Title: Response Patterns to the Electric Stimulation of Epidural Catheters in Term Pregnant Women: A Randomized Controlled Trial of Uniport Versus Multiport Catheters.
Brief Title: Response Patterns to the Electric Stimulation of Epidural Catheters in Term Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-05
Record Dates: First submitted 2014-10-09; First posted 2014-10-24 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Labor Pain
Keywords: Tsui Test; Labour; Epidural catheter
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uniport catheter (Active Comparator): 19 gauge uniport epidural catheter
  Interventions: Device: Trans-catheter electric stimulation test
- Multiport catheter (Active Comparator): 19 gauge multiorifice epidural catheter
  Interventions: Device: Trans-catheter electric stimulation test

INTERVENTIONS:
Device: Trans-catheter electric stimulation test
  Other Names: Tsui test

SUMMARY:
Lumbar epidural analgesia is commonly used for labor pain relief due to its effectiveness and safety. Despite its very high success rate, the epidural technique remains a rather blind technique and failures continue to occur. The correct placement of an epidural catheter, however, remains a clinical problem, since there is no imaging technique that could be used at the bedside to determine the exact positioning of the catheter. The technique of a trans-catheter electric stimulation test (TCEST) has been successfully used to detect the proper epidural catheter location for pediatric, post-operative and laboring obstetric patients. The response to the TCEST with the uniport (single hole) epidural catheters has been well described. There is a growing body of evidence that multiport epidural catheters provide an advantage to uniport catheters, since additional ports likely allow for an enhanced distribution of the local anesthetic solution. This was shown to result in a lower incidence of inadequate analgesia, including unilateral sensory blockade and missed sensory segments. The characteristics of the TCEST response using a multiport catheter remain to be determined. The aim of this study is to compare the response patterns to the TCEST using a single port versus multiport wire reinforced epidural catheters. The hypothesis of this study is that the incidence of a bilateral response to the TCEST will be higher in the multiport catheter as compared to the uniport catheter.

DETAILED DESCRIPTION:
This will be a randomized double-blind controlled study. After recruitment of the patient, epidural anesthesia will be performed in the standard fashion employed in the investigators institution by a resident, fellow, or staff. Spinal ultrasound will be used prior to performing the epidural catheter insertion. Patients will be randomly allocated into two different groups to receive either a 19 gauge uniport catheter or a 19 gauge multiorifice catheter (Arrow Flextip plus, Arrow International Inc., Reading, PA). After securement of the catheter, the TCEST will be performed. The test will be repeated at 5 minutes, following a test dose, to determine the change in intensity of current required to elicit the motor response. Following the second testing, a loading dose of the standard anesthetic solution will be administered. The sensory level to ice will be tested at 20 minutes following injection of the loading dose of bupivacaine and fentanyl. The sensory level will be assessed from the sacral to the thoracic levels, bilaterally Failure of the epidural analgesia will be assessed, defined as no evidence of a sensory block to ice and absent pain relief. The need for catheter replacement will be determined within 2 hours of the completion of the loading dose.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age requesting an epidural for labor and delivery
* Able to communicate in English
* Informed consent

Exclusion Criteria:

* Refusal to provide written informed consent
* Unable to communicate in English
* Allergy or hypersensitivity to lidocaine, bupivacaine or fentanyl
* Abnormal vertebral anatomy, including previous spine surgery and scoliosis
* Coexisting neurological disorders
* Implanted electronic devices

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Motor response pattern | 5 minutes
  Motor response pattern to the electrical stimulation of the epidural catheter, either unilateral or bilateral

SECONDARY OUTCOMES:
Current (mA) | 5 minutes
  The current (mA) needed to elicit a motor response at control and at 5 minutes after the test dose
Sensory level | 20 minutes
  The sensory level to ice at 20 minutes following injection of the standard epidural loading dose. The sensory level will be assessed from the sacral to the thoracic levels, bilaterally
Epidural block failure | 20 minutes
  Failure of the epidural analgesia, defined as no evidence of a sensory block to ice and absent pain relief
Catheter replacement | 2 hours
  Need for catheter replacement within 2 hours of the completion of the loading dose

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada